CLINICAL TRIAL: NCT00348218
Title: Pilot Study To Evaluate The Efficacy Of Neurovision'S NVC™- Vision Correction Technology For The Improvement In Visual Acuity In Myopic Children And Slowing Down Of Myopia Progression
Brief Title: Pilot Study of Neurovision to Improve Vision and Slow Myopia Progression in Children With Myopia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: NeuroVision (Industry); Health Promotion Board, Singapore (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R462/11/2006
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Myopia
Keywords: Neurovision; Myopia Therapy
MeSH Terms: conditions — Myopia

INTERVENTIONS:
Device: NeuroVision

SUMMARY:
This is a pilot study to assess the effectiveness of Neurovision treatment in the improvement of vision in children being under-corrected and to assess the effectiveness of Neurovision treatment in slowing down myopia progression in children.

DETAILED DESCRIPTION:
NeuroVision's NVC vision correction technology is a non-invasive, patient-specific computerized treatment based on visual stimulation and facilitation of neural connections responsible for vision. NeuroVision's Neural Vision Correction TM (NVC) technology has been developed through research focused solely on optimizing performance of the neural or "back end" of the visual system, and is based on two decades of visual neuroscience research by the founder, Dr Uri Polat, whose work, which has been published in leading scientific journals, relates to understanding how the brain processes visual information, how neural activity is related to visual perception, and how visual processing interacts with other neural systems.

The technology has been clinically proven in the treatment of adult amblyopia, which until now has been considered untreatable, with a RCT in which follow-up of up to 2 years shows good retention of visual improvement. The company has received FDA 510(k) marketing clearance indicating NVC for the treatment of adult amblyopia in patients 9 years or older in the US. The company also received a Medical CE-Mark to market its Amblyopia and Low-Myopia products in the European Union. Company products are also approved for use in Israel by the Israeli Ministry of Health - Device License Authority. Additional proof-of-concept studies have been performed in Israel and Singapore indicating the technology's potential to improve vision of subjects having low myopia.

Today, NeuroVision commercially offers the Low Myopia treatment in Singapore. Initial results of the commercial treatment are even better than the proof-of-concept studies, emphasizing the importance of patient motivation and compliance in this treatment.

Based on the promising results of the Low Myopia treatment in adults, this study intends to evaluate the efficacy of NVC treatment in myopic children, by improving their quality of vision and reducing the progress rate of their Myopia.

The first objective of this study is to evaluate the improvement of visual acuity in children being under-corrected. As the myopia increases rapidly in many children, their habitual eyewear cannot match their exact degree of myopia on a day by day basis. As a result, many children suffer from reduced quality of vision (as shown also in data from the Singapore Cohort Study of the Risk Factors of Myopia [SCORM] study). Therefore, the first goal of this study is to evaluate the effectiveness of NeuroVision treatment in the improvement of the under-corrected visual acuity of these children.

The second objective is to evaluate the effectiveness of NeuroVision treatment in the reduction of the myopia progression rate in children. As detailed later on in this document, studies on animals showed that under-correcting myopia can reduce its progression rate (or even result in emmetropization). Therefore, the second goal of this study is to evaluate the possibility of significantly under-correcting myopia in children that had undergone NeuroVision treatment, and check how it affects the progression of their myopia.

To achieve the above objectives, a large scale (few hundred subjects) clinical study on school children, is required. This pilot study is designed to examine the feasibility of such a large scale study, from clinical, administrative and logistic points of view.

Treatment flow and process

The treatment flow is composed of the following phases

1. Screening and Enrollment

   The Screening Evaluation phase includes the following steps:
   1. Demographic details
   2. General medical history
   3. Baseline Examination I. Manifest Subjective and Objective refraction II. Accommodation amplitude, PRA and NRA III. Distance visual acuity (Monocular and binocular Under-corrected Visual Acuity, and Best Corrected Visual Acuity - BCVA) IV. Cycloplegic Objective and Subjective refraction V. Distance cycloplegic under-corrected visual acuity. VI. Ocular axial length measurements

   For detailed description of the above examinations, refer to Appendices A-B.

   After the completion of all the required examinations, subject's data will be reviewed and study investigators make a final enrolment decision.

   Before starting the computerized evaluations, subjects will undergo an additional Distance Visual Acuity and Contrast Sensitivity examinations at the school.

   The results of these additional examinations will be used as a baseline reference for the periodic examinations that will be done during the treatment period.

   Enrolled Subjects will be requested to complete a QOV/QOL Questionnaire 1 (Annex E) before the treatment starts
2. NVC Computerized Evaluation

   The Computerized Evaluation sessions are conducted in order to allow the NVC system to identify the visual abilities and inefficiencies and to thereby define individual parameters that will affect the subject's treatment plan.

   This phase is comprised of two (2) to three (3) sessions.

   Training Glasses:

   NeuroVision will determine the power of the training eyeglasses the subject will need for the NVC treatment start. The possible training glasses are 0.5DS, 1.0DS or 1.5DS less than the subject's full prescription. In some cases, there will be no training glasses.

   In some cases a subject might be instructed to train one eye only for a part of the treatment sessions. The other eye will be then covered by a semi-translucent lens.

   The decisions are made by NeuroVision based on the subject's best refractive correction, his/her under-corrected VA and the computerized evaluation, and will be reported to the study coordinator.
3. NVC Treatment

   The total number of sessions to complete the treatment course is not defined in advance. It is determined by the NVC system during the course of treatment according to each subject's visual abilities and performance. Typically patient should undergo 30 sessions during this phase.

   The subject should perform on average three (3) sessions per week.

   During this phase no visit interruptions longer than two (2) weeks on aggregate are permitted.

   Periodic visual acuity and contrast sensitivity examinations should be performed after every 5 treatment sessions in the school

   As progress is made, the training glasses previously provided to the subject may be replaced by other training glasses with less power, or entirely removed. The clinician and the subject will be informed about the training glass replacement in advance.

   After completing 15 treatment sessions (mid-term), subjects will be requested to complete a QOV/QOL Questionnaire 2 (Annex F) before commencing Treatment Session 16.

   NOTE:

   WHEN VA TEST AND THE TREATMENT SESSION ARE TO BE PERFORMED AT THE SAME VISIT, PERIODIC VA TESTS SHOULD BE ALWAYS CONDUCTED BEFORE THE PERFORMANCE OF A TREATMENT SESSION!
4. End of Treatment Decision

   Subject will terminate the treatment sequence according to the end of treatment criteria (see summary of study design)

   Following the end of Treatment decision, the subject should be scheduled for Post Treatment Examinations (PTE) within 2 weeks.

   For follow up visits, visit range allowed is within +/- two weeks of the expected dates
5. Post Treatment Examination (PTE)

   The Post Treatment Examination at SERI will include visual acuity tests, amplitude of accommodation, relative accommodation, cover test, cycloplegic refraction and distance under-corrected visual acuity and axial length measurement.

   Subjects will be requested to complete a QOV/QOL Questionnaire 2 (Annex F)
6. Prescription of under-corrected eyewear

   After the end of the treatment, subjects should be prescribed with under-corrected eyewear.

   The under-corrected eyewear should be the lowest possible refractive correction in which that subject has at least 6/12 (0.3 LogMAR) binocular VA.

   The subject should be instructed to use the new eyewear instead of the current one (if any) for at least the 12 months monitoring period.
7. Follow-Up Examinations at Months 3, 6, 9 and 12

Follow-Up Examinations at Months 3, 6, 9 and 12 post treatment at SERI will include visual acuity tests, amplitude of accommodation, relative accommodation, cover test, cycloplegic refraction and distance under-corrected visual acuity.

In case that the subject's binocular VA with the under-corrected eyewear is worse than 6/12 (0.3 LogMAR) for 2 consecutive follow-up visits, new eyewear should be prescribed to allow at least 6/12 binocular VA.

At Follow up Month 6 and 12, subjects will be requested to complete a QOV/QOL Questionnaire 2 (Annex F)."

ELIGIBILITY:
Inclusion Criteria:

1. The subject's age is between 7 to 9 years.
2. The subject's cycloplegic refraction is at least -1.0DS in either eye.
3. The subject's manifest spherical equivalence does not differ by more than 1.0 D from cycloplegic spherical equivalence
4. The subject's visual acuity with an under correction of 1DS (compared to the manifest subjective VA), in both eyes, should not exceed 0.6 LogMAR.
5. The subject's best corrected visual acuity 0.04 LogMAR (either eye)
6. The subject is cognitively intact and is able to follow multiple step instructions.
7. The subject and his parents/legal guardians are very keen to improve the habitual visual acuity and to reduce the progression rate of myopia
8. The subject is able and willing to attend all study sessions and visits at the required frequency:

   * The total number of treatments is individual, approximately 30 and no more than 40.
   * The required pace for the treatment sessions is at least 3 sessions per week.
   * No foreseen interruptions longer than 2 weeks during the treatment course.
9. The subject is able to cease contact lens wear from Baseline examination onwards until the end of the treatment period (phase I).
10. The subject's parent/legal guardian agrees to sign the Informed Consent Form (See Appendix D)
11. Subject's parent/legal guardian agrees to follow the study instruction including use of optical aids

Exclusion Criteria:

1. The subject suffers from any other eye disease(s) or other causes for the reduced visual acuity, aside from myopia and/or astigmatism.
2. The subject suffers from myopia-related visual complications resulting in visual loss, including myopic macular degeneration, myopic cataract and previous or pre-existing myopic retinal detachment.
3. The subject is suffering from Diabetes Mellitus.
4. The subject suffers from binocular vision problems, such as high exophoria / divergent squint / nystagmus
5. The subject has an activity limitation due to medical disorders (including migraines, seizure disorders, etc.), medications, or emotional status that might potentially impair the subject's ability to perform the treatment.

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2006-06; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Manifest Subjective and Objective refraction
Accommodation amplitude, PRA and NRA
Distance visual acuity (Monocular and binocular Under-corrected Visual Acuity, and Best Corrected Visual Acuity - BCVA)
Cycloplegic Objective and Subjective refraction
Distance cycloplegic under-corrected visual acuity.
Contrast Sensitivity
Ocular axial length measurements

CONTACTS AND LOCATIONS:
Overall Officials: Donald Tan, FRCS, Principal Investigator — Singapore Eye Research Institute; Wei Han Chua, FRCS, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore

REFERENCES:
- [Background] Polat U, Ma-Naim T, Belkin M, Sagi D. Improving vision in adult amblyopia by perceptual learning. Proc Natl Acad Sci U S A. 2004 Apr 27;101(17):6692-7. doi: 10.1073/pnas.0401200101. Epub 2004 Apr 19. PMID 15096608
- [Background] Lim KL, Fam HB. NeuroVision treatment for low myopia following LASIK regression. J Refract Surg. 2006 Apr;22(4):406-8. doi: 10.3928/1081-597X-20060401-20. PMID 16629076
- [Background] Polat U, Mizobe K, Pettet MW, Kasamatsu T, Norcia AM. Collinear stimuli regulate visual responses depending on cell's contrast threshold. Nature. 1998 Feb 5;391(6667):580-4. doi: 10.1038/35372. PMID 9468134
- [Background] Levi DM, Polat U, Hu YS. Improvement in Vernier acuity in adults with amblyopia. Practice makes better. Invest Ophthalmol Vis Sci. 1997 Jul;38(8):1493-510. PMID 9224277
- [Background] Polat U, Norcia AM. Neurophysiological evidence for contrast dependent long-range facilitation and suppression in the human visual cortex. Vision Res. 1996 Jul;36(14):2099-109. doi: 10.1016/0042-6989(95)00281-2. PMID 8776476
- [Background] Sagi D, Tanne D. Perceptual learning: learning to see. Curr Opin Neurobiol. 1994 Apr;4(2):195-9. doi: 10.1016/0959-4388(94)90072-8. PMID 8038576
- [Background] Polat U, Sagi D. Spatial interactions in human vision: from near to far via experience-dependent cascades of connections. Proc Natl Acad Sci U S A. 1994 Feb 15;91(4):1206-9. doi: 10.1073/pnas.91.4.1206. PMID 8108388
- [Background] Polat U, Sagi D. Lateral interactions between spatial channels: suppression and facilitation revealed by lateral masking experiments. Vision Res. 1993 May;33(7):993-9. doi: 10.1016/0042-6989(93)90081-7. PMID 8506641
- See also: Singapore Eye Research Institute Website — http://www.seri.com.sg/